CLINICAL TRIAL: NCT03645616
Title: Reliability of Functional Tests for Individuals With Chronic Low Back Pain.
Brief Title: Reliability of Function Tests for People With Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alessandro Haupenthal (Other)
Collaborators: Santa Catarina Federal University (Other)
Responsible Party: Sponsor-Investigator, Alessandro Haupenthal, Principal Investigator, Universidade Federal de Santa Catarina
Organization: Universidade Federal de Santa Catarina (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2.537.100
Record Dates: First submitted 2018-08-20; First posted 2018-08-24 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Low Back Pain; Adult
Keywords: Musculoskeletal disease; Stress test; Reproducibility; Gait Speed
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Diseases | interventions — Walk Test

STUDY DESIGN:
Masking Description: All data were color coded to guarantee that the investigator who processed the data was blinded to the conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Tests (Experimental): Participants undertook 6-minute walk test, 10 meters walk test and 30 second sit to stand test.
  Interventions: Diagnostic Test: 6-minute walk test; Diagnostic Test: 10 meters walk test; Diagnostic Test: 30 Second Sit to Stand Test

INTERVENTIONS:
Diagnostic Test: 6-minute walk test — First day: Participants undertook 6-minute walk test. There was a 30-minute interval between the first and second test, when the patient was asked to rest. During the resting period, they respond a pain intensity, functional capacity and physical activity level questionnaire.
  Second day: the participants repeated the test and questionnaires.
Diagnostic Test: 10 meters walk test — First day: After the second 6-minute walk test the participants perform the 10-meter walk test, the test must be performed three times with a 30-second interval, at the end the average test velocity.
  Second day: the participants repeated the test.
Diagnostic Test: 30 Second Sit to Stand Test — At the end of the tests the participants perform the 30 Second Sit to Stand Test on the first and second day.

SUMMARY:
Back pain is often accompanied by changes in function. The performance of individuals with their backs on their wills may become more functional. It is believed that the test will present good to excellent reliability in individuals with chronic back pain. From this, it can be used in the clinic to verify the functional capacity of these individuals.

DETAILED DESCRIPTION:
This study will be performed to verify the reliability of the functional tests for individuals with back pain. A study in which individuals with back pain will be assessed on the first day and after the interval of seven days. They should perform the 6-minute walk test and answer some questionnaires such as the Roland Morris - disability questionnaire, the IPAQ - physical activity level questionnaire and Numeric Rating Scale, after the tests will be performed Timed 10-Meter Walk Test and 30 Second Sit to Stand Test. To avoid a random error, a minimum sample size of 30 participants is required. For statistical analysis, Shapiro-Wilk test will be used for data normalization and the reliability between measurements will be calculated through do Intraclass Correlation Coefficients, standard error of measurement and Minimal Detectable Change. There were no studies in the literature and recorded in the Clinical Trials that evaluated the reliability of these tests for individuals with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes aged 20 to 65 years and low back pain for more than 3 months.

Exclusion Criteria:

* Acute pain of back pain that disables the performance of the tests.
* Pregnancy.
* Neoplasms.
* Known heart, lung or metabolic diseases.
* Hypotension (BP < 90 x 60 mmHg) or stage II hypertension (BP > 140 x 90 mmHg), medicated or not.
* Fall or faint in the previous two months.
* Have not undergone any spinal surgery.
* Have not had neuromuscular impairment in the last three months and who need help to follow the instructions.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Distance traveled in meters. | The individual will perform 42 minutes of testing, two walking tests of 6 minutes plus 30 minutes of rest
  Measured by the 6-minute walk test. Individuals should walk in a 30 meter corridor for 6 uninterrupted minutes.

SECONDARY OUTCOMES:
Pain intensity | 5 minutes
  Measured through the Numerical Rating Scale, being considered an improvement of pain, the reduction of 2,5 points in the NRS. Evaluated at the beginning and after the tests.
Functional Incapacity | 10 minutes
  Measured using the Roland Morris functional disability questionnaire considering improvement the decrease of 2.5 points.
Physical activity level | 10 minutes
  The scores obtained through the International Physical Activity Questionnaire (IPAQ) are obtained through the minutes of activities performed per week, classifying the individual as very active, active, irregularly active and sedentary
Gait Speed | 5 minutes
  Measured through the 10 meters walk test that measures walking speed in meters per second for a short period. Individual walks without assistance 10 meters (32.8 feet) and the time is measured for the intermediate 6 meters (19.7 feet) to allow for acceleration and deceleration.
Functional lower extremity strength | 30 seconds.
  Measured through the 30 Second Sit to Stand Test, which evaluates the functional limb strength with the number of sit and stand repetitions for 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Aline L Ballico, Student, Principal Investigator — Santa Catarina Federal University
Locations (1):
- Santa Catarina Federal University, Araranguá, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Britto RR, Sousa LAP. Teste de caminhada de seis minutos- Uma normatização brasileira. Fisioterapia em Movimento 19(4):49-54, 2006.
- [Background] Chou R, Deyo R, Friedly J, Skelly A, Hashimoto R, Weimer M, Fu R, Dana T, Kraegel P, Griffin J, Grusing S, Brodt ED. Nonpharmacologic Therapies for Low Back Pain: A Systematic Review for an American College of Physicians Clinical Practice Guideline. Ann Intern Med. 2017 Apr 4;166(7):493-505. doi: 10.7326/M16-2459. Epub 2017 Feb 14. PMID 28192793
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520
- [Background] Lamoth CJ, Meijer OG, Daffertshofer A, Wuisman PI, Beek PJ. Effects of chronic low back pain on trunk coordination and back muscle activity during walking: changes in motor control. Eur Spine J. 2006 Jan;15(1):23-40. doi: 10.1007/s00586-004-0825-y. Epub 2005 Apr 29. PMID 15864670